CLINICAL TRIAL: NCT00561587
Title: Quetiapine vs. Placebo in Alcohol Relapse Prevention - a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Prof. Ursula Havemann-Reinecke, MD PhD, Department of Psychiatry and Psychotherapy, GEORG-AUGUST-UNIVERSITY GÖTTINGEN, GERMANY
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 87, 1, 2007_01_30
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2008-01

CONDITIONS: Alcohol Relapse Prevention; Alcoholism; Alcohol Drinking; Alcohol Consumption; Alcohol Abuse
Keywords: novel antipsychotic; quetiapine; depression; psychopathology
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Seroquel®
- 2 (No Intervention)

INTERVENTIONS:
Drug: Seroquel® — dosage form: oral, adjusted in the range of 25 to max. 300 mg /day
  Other Names: Quetiapine
  Arms: 1

SUMMARY:
Due to Quetiapine's particulars and the promising receptor profile, we want to examine the efficacy concerning relapse prevention of alcoholics suffering from persisting craving and/or affective symptoms (persisting sleep disorder, persisting excitement, persisting depressive symptoms, persisting anxiety symptoms) in comparison to matching placebo in a double-blind pilot study.

We further want to compare the course of the above mentioned craving and affective symptoms under medication with quetiapine / matching placebo.

DETAILED DESCRIPTION:
Naltrexone and Acamprosate are the best evaluated and established therapy options in relapse prevention of alcoholics at present (Litten et al. 1996, Mann et al. 2004). Studies on cue exposure showed that Naltrexone (Monti et al. 1999) and Haloperidol (Modell et al. 1993) block stimuli triggered craving. In addition, they indicate that both may also stop the craving for further alcohol consumption that is induced by a priming dose of alcohol (Modell et al. 1993). However, the clinical relevance of Haloperidol is rather limited due to the risk of extrapyramidal side effects. New atypical dopamine antagonists are reported to have this profile as well, but without the risk of developing extrapyramidal side effects. In a placebo-controlled clinical trial, the atypical antipsychotic Olanzapine has proved to reduce craving for alcohol both after alcohol exposure and a priming dose of alcohol in non-dependent heavy social drinkers (Hutchison et al. 2001). However, Amisulpride in a dose of 50 mg per day failed to prevent alcohol relapse in a double-blind, placebo-controlled study in 71 patients over 6 months (Marra et al. 2002).

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence according to ICD-10 and DSM-IV since a minimum of 12 months.
* Detoxified male or female aged between 18 and 65 years.
* Abstinence for a minimum of 7 days and maximum of 21 days before randomization.
* Craving : minimum of 5 points at randomisation (OCDS-G)
* Free informed consent has been given in written form.
* Women of childbearing potential must use a medically accepted method of contraception.

Only methods with a Pearl-index lower than 1% are regarded as acceptable such as hormonal contraception, surgical sterilization, bilateral ovarectomy, and postmenopause (WHO definition: natural menopause retrospectively for at least one year amenorrhoe) without hormonal replacement therapy within the past 5 months.

Exclusion Criteria:

* Patients suffering from psychotic diseases and/or depression with psychotic symptoms and/or demented patients, patients with longlasting continous treatment with psychotropic drugs.
* Known substance abuse other than alcohol or nicotine (except dependence in full remission) as defined by DSM-IV criteria. Patients with a positive urine toxicology screen will be excluded only if they satisfy the DSM-IV criteria for abuse or dependence.
* Hepatitis (GGT or AST three times above normal range).
* An absolute neutrophil count (ANC) of ≤ 1.5 x 109 per liter.
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

unstable DM defined as enrollment glycosylated hemoglobin (HbA1c)>8.5 %; patients admitted to hospital for treatment of DM or DM related illness in past 12 weeks; patients not under physicians care for DM; physicians responsible for patient´s DM care has not indicated that patient´s DM is controlled; physician responsible for patient´s DM care has not approved patient´s participation in the study; patient has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to randomization. [For thiazolidinediones (glitazones) this period should not be less than 8 weeks]; patients taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks.

Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.

Evidence of clinical relevant disease or clinical finding that is unstable or that, in the opinion of the investigator, would be negatively affected by study medication or that would affect study medication.

* Patients who, in the investigator's judgment, pose a current serious suicidal risk or have made a suicide attempt within the past 6 months.
* Restricted or complete legal incapacity.
* Additional psychotherapy 1 month prior to randomisation or during participation in the study.
* History of idiopathic orthostatic hypotension, or condition that would predispose to hypotension (e.g. dehydration, hypovolemia).
* Risk of transmitting human immunodeficiency virus (HIV) or hepatitis B, C, via blood or other body fluids (as judged by the investigator). Positive HIV-serology in the screening visit.
* Known regular treatment with Quetiapine prior to randomisation.
* Hypersensitivity to Quetiapine or other constituents of the investigational product.
* Simultaneous intake of Cytochrome-P-450-3A4- inducers or inhibitors: Use of drugs that induce or inhibit the hepatic metabolizing cytochrome 3A4 enzymes within 2 weeks prior to randomization or during the study period, e.g. the inducers: carbamazepine, phenytoin, barbiturates, rifampicin, rifabutin, glucocorticoids, thioridazine and St. Johns wort, and e.g. the inhibitors: HIV-protease-inhibitors, antimycotics of the azole type (e.g. ketoconazole (except for topical use), itroconazole, fluconazole), erythromycin, clarithromycin, fluvoxamine, nefazodone, troleandomycin, indinavir, nelfinavir, ritonavir, and saquinavir
* Female patients who are pregnant or are lactating. Women of childbearing potential not using a medically accepted method of contraception with a Pearl-index > 1%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
1) blood alcohol concentration > 1.0 per mille 2) alcohol consumption > 40 g/day (females) or > 60 g/day (males) 3) continuous intake of alcohol during more than 5 consecutive days (independent of the amount of alcohol) | 7 month

SECONDARY OUTCOMES:
first consumption of any ethanol,number of drinking and abstinence days,craving measured by the total score of the OCDS-G,STAI,PSQI,depression measured with MADRS and BDI,Amount of total daily cigarette consumption,FTND,CO-breath analysis variance | 7 month

CONTACTS AND LOCATIONS:
Overall Officials: Karl Mann, MD PhD, Principal Investigator — Dept. of Addictive Behavior and Addiction Medicine, Central Institute of Mental Health, Mannheim, University of Heidelberg, Germany; Bernhard Croissant, MD PhD, Principal Investigator — Dept. of Psychiatry and Psychotherapy, Hospital Sigmaringen, University of Tuebingen; Ursula Havemann-Reinecke, MD PhD, Study Director — Department of Psychiatry and Psychotherapy, Georg-August-University, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Goettingen, Göttingen, Lower Saxony, Germany